CLINICAL TRIAL: NCT02315222
Title: Impact of Dietary Supplements on Oral and Periodontal Wound Healing
Brief Title: Dietary Supplements and Periodontal Wound Healing
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Milan (Other)
Responsible Party: Principal Investigator, Giulio Rasperini, Professor, University of Milan
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Regenium
Record Dates: First submitted 2014-12-09; First posted 2014-12-11 (Estimated); Last update posted 2014-12-11 (Estimated); Status verified 2014-12

CONDITIONS: Periodontitis
Keywords: Nutriomics; Dietary supplements; Scaling and root planing; full mouth disinfection
MeSH Terms: conditions — Periodontitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Test (Active Comparator): Dietary Supplementation
  Interventions: Dietary Supplement: Regenium; Procedure: Full Mouth Disinfection
- Control (Placebo Comparator): Placebo Supplementation
  Interventions: Dietary Supplement: Placebo; Procedure: Full Mouth Disinfection

INTERVENTIONS:
Dietary Supplement: Regenium
  Arms: Test
Dietary Supplement: Placebo
  Arms: Control
Procedure: Full Mouth Disinfection

SUMMARY:
Patient with periodontal disease undergoing full mouth disinfection will be given dietary supplements or placebo and reevaluated after 3 months.

DETAILED DESCRIPTION:
Introduction The beneficial effect of vitamins and dietary supplements on oral wound healing has been recently reported in clinical trials (for review see Van der Valden, JCP 2011). In periodontal tissue, the imbalanced ratio between virulence of pathogens bacteria and proportionate host response induce a destructive process of periodontal ligament, cementum and alveolar bone. The importance of micronutrients including vitamins, calcium and antioxidant for periodontal health was reported in several clinical studies and the integration between traditional (non surgical and surgical interventions) and micronutritional approaches were proposed for treatment of periodontitis (Van der Velden et al. 2011).

Clinical trials reported that daily supplement of fruit, vegetable and berry juice powder, vitamin D, Calcium seems to improve periodontal health in patients with chronic periodontitis that were treated with non-surgical or surgical periodontal therapy or were in maintenance program (Chapple et al 2012, Garcia et al 2011, Miley et al 2009, Bashutski et al. 2011). However, the beneficial effects of micronutrients on periodontal health and healing need to be more deeply investigated. Furthermore, a dietary supplement specifically formulated for periodontal health needs to be tested.

Regenium is a dietary supplement with Q-TER (coenzyme q10 terclatrate), DHA Omega 3, Boswellia serrata, Vitamins and mineral salts that was formulated to improve the collagen formation and the maintenance of the health of oral mucosa. Q-TER plays a key role in the ATP synthesis and energetic metabolism, and has a strong antioxidant function. A recent study also reported the function of Q-10 as inhibitor of osteoclast differentiation (Moon et al. 2012). DHA Omega 3 (Resolvine) has an important antioxidant function, affecting the cellular aging and moderates the anti-inflammatory mechanisms. Boswellia serrata showed beneficial effects on wound healing and contraction (Mallik et al. 2010). This micronutrient reduces the synthesis of leukotrienes in intact neutrophils by inhibiting 5-lipoxygenase, the key enzyme involved in the biosynthesis of leukotrienes and in the inflammatory process.

The aim of the present study is to evaluate if patients affected by severe periodontal disease and treated with periodontal non-surgical therapy benefit from dietary supplements (Regenium). It will be assessed the effect of Regenium on clinical parameters of periodontal wound healing and on systemic inflammation related to periodontal disease.

1. Experimental procedure

   1.1 Study population A total of 60 patients afflicted with severe periodontal disease and that need for non-surgical periodontal therapy will be enrolled.

   Inclusion criteria
   * severe periodontal disease: at least 2 sites with Probing Pocket Depth (PPD)>7mm, Bleeding On Probing (BOP)> 25%
   * Age between 18 and 65 years
   * Signed informed consent

   Exclusion criteria:
   * Systemic diseases that may affect periodontal status
   * Metabolic disorders
   * Nutritional conditions that may alter the formation and maturation of connective tissue
   * Pregnancy or lactation

   1.2 Subject protection Informed consent will be obtained from all subjects to be entered in the study. In obtaining the informed consent and in the conduct of the study the principles outlined in the Declaration of Helsinki on experimentation involving human subjects should be adhered to. At each visit, the clinician will evaluate patients for any untoward effects. In case a patient requires any treatment during the course of the study, the necessary treatment will be provided at the discretion of the clinician and according to the current standard of care.

   1.3 Treatment After including patient in the study, each patient will be randomly assigned to one of the experimental groups (test, control). At T0 clinical measurements will be harvested, saliva samples will be collected and serum analysis will be performed. Furthermore each patient will receive oral hygiene instructions and regular professional supragingival debridement. Therapy with Regenium or placebo will be given to the patient and will start at T0.

   Four weeks after starting the therapy (T1), clinical measurements and saliva samples will be harvested and serum analysis will be performed. After measurements the one-stage full-mouth disinfection will be performed as following described. Scaling and root planing of all pockets will be performed within 24 h in combination with an extensive application of chlorhexidine (0.20%) to all intra-oral niches such (periodontal pockets, tongue dorsum, tonsils) and in combination with systemic antibiotic treatment (amoxicillin cp. 1gr 2/die + 250 mg metronidazole 3/die).

   To resume patients will intake Ragenium or placebo for 3 months (from 1 months before and until 2 months after non surgical periodontal therapy), each patient will intake one pill of Regenium Tablet in the morning (with breakfast) and one capsule of Regenium Capsule in the evening (with dinner). Patients assigned to the control group (n=30) will intake placebo tablets and capsules as prescribed in the test group. Compliance will be evaluated by pill counting at the end of the study.

   Three months after therapy with Regenium or placebo (T2), clinical measurements and saliva samples will be harvested and serum analysis will be performed.

   Treatment assignment To enter a patient into the study each investigator will fill in a screening and an entry form and fax them to the Central Registrar located at the Clinical Research support Unit of Periodontology, Dental Clinic, Dep. of Biological, Surgical and Dental Sciences, University of Milan, Fondazione IRCCS Ca' Granda Polyclinic Milan, Italy. Following receipt of these forms, the Registrar will proceed to verify satisfaction of all entry criteria and will enter the subject into the study. Patient codes will be assigned consecutively and will be made of a total of 2 digits that will encode the subject number (from 01 to 60). These will be assigned at the first visit, verifying the inclusion criteria and entering the patient into the study. After having been entered patients into the study, experimental patients will be randomly assigned by Central Registrar to one of the two treatment regimens according to pre-defined randomization tables.

   A balanced random permuted block approach will be used to prepare the randomization tables in order to avoid unequal balance between 2 treatments. In order to reduce the chance of unfavorable splits between test and control patients in terms of key prognostic factors, the randomization process will take into account the following variable: smoke. Treatment assignment will be noted in the registration and treatment assignment form that will be kept by the central registrar. To conceal assignment from the investigator until the time, at the end of the non-surgical periodontal therapy the central registrar will instruct the investigator to assign a sealed envelope containing the treatment for each patient, every envelop is endowed of a Treatment's Code, composed by a letter (that corresponds to the clinical center) and two numbers.

   When a patient enters in the study the investigator assigned him a sequential Patient's Code, than the clinician sends Screening Form and Entry Form to the study registrar. The central registrar will match the randomization envelope with the subject number based on the randomization tables and he send the Registration Form, with the correspondence between Patient's Code and Treatment's Code. Following receipt of the registration form from the Central Registrar, the investigator will prescribe the treatment (Regenium or placebo) to the patient and will book all the subsequent appointments according to the protocol.
2. Measurements Clinical measurements To evaluate the inflammatory status, plaque control and severity of periodontal disease, clinical measurements will be taken at T0 (immediately before starting with dietary supplements or placebo), at T1 (4 weeks after starting supplementation) and at the last day of supplementation (T2= 3 months after T0).

The following clinical parameters will be taken:

* Full Mouth Plaque Score (FMPS), Full Mouth Bleeding Score (FMBS)
* Periodontal Pocket Depth (PPD), Clinical Attachment Level (CAL), tooth mobility.

All clinical measurements will be taken by a blind calibrated examiner.

Radiographic evaluations An X-Ray status with a parallel technique will be taken at the baseline during the diagnostic process of periodontal disease.

Serum analysis

Blood test will be performed at T0, T1 and T2 in all patients to evaluate the systemic inflammation and to assess changes on this condition after periodontal treatment and dietary supplements intake. The following blood markers of systemic inflammation will be evaluated (Graziani et al. 2010):

* High sensitivity C reactive protein (hsCRP)
* D-dimers and renal function (cystatin C)

Whole Saliva Collection Unstimulated whole saliva will be collected from each subject at the beginning of the appointment, as previously described by Ramseier et al. Subjects' will vigorously rinsed their mouth with tap water for 20 seconds in order to remove gross debris. The subject then expectorates the water. Following a waiting period of 2 minutes, subjects will tip their head over the graduated test tube and passively expectorated whole saliva into the plastic funnel placed inside the plastic tube (Mandel et al. 1976). Each tube will be labeled with the subject's initials, harvest date and sample name. The collection will be completed once 2mL of whole saliva is collected, or a maximum of 15 minutes of sampling time is reached. The sample will then immediately placed on ice, supplemented with a proteinase inhibitor combination of 1% aprotinin (1mg/ml) and 0.5% phenylmethylsulphonyl fluoride (PMSF) (200mM in MeOH) (Sigma Chemical Company, St-Louis, MO), and aliquotted prior to storage at -20°C until analysis.

Salivary Biomarkers Analysis Inflammatory biomarkers expression will be quantified using a custom human cytokine protein array|| for the evaluation of matrix metalloproteinase-8 and -9 (MMPs-8 and -9).

Upon receipt, the Quantibody® Array kits will be stored at -20°C. Prior to each assay, whole saliva samples will be thawed at room temperature and microcentrifuged for 5 minutes to obtain a cell-free supernatant for analysis.

Each slide containing cytokine standards used for making known serial dilutions, with sample diluent serving as the negative control, and experimental samples will then be incubated overnight at 4°C followed by washing unbound materials. The detection antibody will then bound to the antigens within each well. Cy3 equivalent dye-conjugated streptavidin will be pipetted in each well, which binds to the detection antibody associated with immune complexes. The slides will be incubated and covered with aluminum foil to avoid light exposure and the fluorescence from each well was detected using a laser scanner.¶ The resultant signals of the samples will be compared to the standard curve for each of the cytokines in order to determine the concentrations of each cytokine within the samples. Data will be extracted and analyzed using microarray analysis software.#

Compliance and its evaluation Compliance is a serious problem for clinical trials, to improve this fundamental aspect of the study, the clinicians will adopt some useful technique.

Every patient will be instructed to download on his smartphone an application that will remind him to take Regenium in the morning and in the evening; secondly the clinician will call the patients two weeks after T0 and two and five weeks after T1, with the pretext to remind the next appointment and to have information about their oral health, but with the real intention to remember and to verify the regular assumption of Regenium. Lastly, at T2, patients will have to bring back the blister, also the empty ones, for the pill counting.

It is important not to say the patients about the pill count, in order to avoid the risk of bias created by patient who throw away the remaining pill the day before the control. To have the blister back, clinicians will say the patients to return blister for wasting reasons, for both package and pills.

References

J.D. Bashutski et al. The impact of vitamin D on periodontal surgery outcomes. Journal of Dental Research, vol 90, pp. 1007-12, 2011.

M. R. Chapple, et al. Adjunctive Daily Supplementation with Encapsulated Fruit, Vegetable and Berry Juice Powder Concentrates and Clinical Periodontal Outcomes: A Double-blind RCT. Journal of Clinical Periodontology, vol. 39, no. 1, pp. 62-72, 2012.

M. N. Garcia, C. F. Hildebolt, D. D. Miley, D. A. Dixon, R. A. Couture, C. L. Spearie, E. M. Langenwalter, W. D. Shannon, E. Deych, C. Mueller, and R. Civitelli, "One-year Effects of Vitamin D and Calcium Supplementation on Chronic Periodontitis,"Journal of Periodontology, vol. 82, no. 1, pp. 25-32, 2011.

F. Graziani, et al. Systemic Inflammation Following Non-surgical and Surgical Periodontal Therapy Journal of Clinical Periodontology, vol. 37, no. 9, pp. 848-54, 2010.

A. Mallik et al. Evaluation of Boswellia Serrata oleo-gum resin for wound healing activity. Der Pharmacia Lettre, , vol. 2, no. 2, pp. 457-463, 2010.

I.D Mandel, and S. Wotman, The salivary secretions in health and disease. Oral Sciences Review, vol 8, pp. 25-47, 1976.

D. D. Miley, M. N. Garcia, C. F. Hildebolt, W. D. Shannon, R. A. Couture, C. L. Anderson Spearie, D. A. Dixon, E. M. Langenwalter, C. Mueller, and R. Civitelli, "Cross-sectional Study of Vitamin D and Calcium Supplementation Effects on Chronic Periodontitis,"Journal of Periodontology, vol. 80, no. 9, pp. 1433-9, 2009.

H. Moon et al., Antioxidants, like coenzyme Q10, selenite, and curcumin, inhibited osteoclast differentiation by suppressing reactive oxygen species generation. Biochemical and Biophysical Research Communications vol. 418, pp. 247-253, 2012.

C.A Ramseier et al., Identification of pathogen and host-response markers correlated with periodontal disease. Journal of Periodontology vol 80, no. 3, p. 436-46, 2009.

U. Van der Velden, D. Kuzmanova, and I. L. C. Chapple, "Micronutritional Approaches to Periodontal Therapy,"Journal of Clinical Periodontology, vol. 38, pp. 142-158, 2011.

ELIGIBILITY:
Inclusion Criteria:

* severe periodontal disease: at least 2 sites with Probing Pocket Depth (PPD)>7mm, Bleeding On Probing (BOP)> 25%
* Age between 18 and 65 years
* Signed informed consent

Exclusion Criteria:

* Systemic diseases that may affect periodontal status
* Metabolic disorders
* Nutritional conditions that may alter the formation and maturation of connective tissue
* Pregnancy or lactation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2014-11; Primary Completion 2015-07 (Estimated)

PRIMARY OUTCOMES:
Clinical Attachment Level (CAL) | 3 months
Periodontal Pocket Depth (PPD) | 3 months

SECONDARY OUTCOMES:
Tooth mobility | 3 months
Full Mouth Bleeding Score (FMBS) | 3 months
Full Mouth Plaque Score (FMPS) | 3 months

CONTACTS AND LOCATIONS:
Locations (3):
- Italy (3):
  - Clinica Odontoiatrica IRCCS Ospedale Maggiore Policlinico, Milan, MI
  - Ospedale Militare, Milan, MI
  - Studio Odontoiatrico Professor Rasperini, Piacenza, PC